CLINICAL TRIAL: NCT03328910
Title: The Relationship Between the Surgical Pleth Index (SPI) and the Postoperative Emergence Delirium in Pediatric Patients After General Anesthesia
Brief Title: The Relationship Between the SPI and the Postop ED
Acronym: SPI_ED
Status: Withdrawn | Type: Observational
Why Stopped: because the instruments for collecting the SPI data from the monitor (S5 collector) could not be imported due to the manufacturer's problem.
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant Professor, Daegu Catholic University Medical Center
Other Study IDs: DCMC#2
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: General Anesthesia
Keywords: Emergence Delirium; pulse oximetry; Children, Preschool
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Analgesia monitoring: After anesthesia induction, all participants received standard anesthesia monitoring, SPI monitor (GE Healthcare, Helsinki, Finland) and bispectral index (BIS). BIS was kept between 40-60, whereas no specific target was determined for SPI. At the end of surgery, anesthesia was terminated and the patients were stimulated to wake up. After the participants were able to breathe spontaneously and obey verbal commands, extubation was carefully performed, and the monitoring of SPI was stopped.
  Interventions: Device: SPI monitor (GE Healthcare, Helsinki, Finland)

INTERVENTIONS:
Device: SPI monitor (GE Healthcare, Helsinki, Finland) — The SPI is derived from pulse rate and pulse wave amplitude measured with photoplethysmography, obtained from the CARESCAPE B650 monitor (GE Healthcare, Finland) with a scale from 1 to 100.

SUMMARY:
Surgical plethysmography index (SPI) is a device that can noninvasively monitor the balance between the nociception and ant-nociception using pulse photoplethysmographic amplitude (PPGA) and heart rate obtained through an oxygen saturation measuring device. SPI has recently been studied as a useful tool to monitor the stress response of patients due to surgery or anesthesia and to guide the appropriate use of analgesics/anesthetics. However, these SPI devices have been developed for adults and have not been studied in pediatric patients with relatively high heart rates, and no direct effects on post-operative arousal excitability have been reported.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 2-7 years with an American Society of Anaesthesiologists physical status (ASA PS) of 1 or 2, who were planned to undergo ophthalmology surgery requiring general anesthesia.

Exclusion Criteria:

* ASA PS 3 or 4
* Presence of developmental delays or neurological diseases
* History of allergies or contraindications to the use of ketamine (increased intracranial pressure, open-globe injury, or a psychiatric or seizure disorder)
* treatment with beta-receptor blockers, beta-receptor agonists or any other drug suspected to interact with the sympathovagal balance
* diseases with impairment of sensitivity (diabetes, polyneuropathy, peripheral arterial obstructive disease et etc)
* pacemaker therapy
* dermal diseases with the affection of the forearm/hand

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 2-7 years with an American Society of Anaesthesiologists physical status (ASA PS) of 1 or 2, who were planned to undergo ophthalmology surgery requiring general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between the SPI during emergence time and the peak emergence delirium score | Observation from approximately 1 hour after the end of operation
  The SPI is attained from waveform finger plethysmography. It is expressed as a numerical index between 0 (total absence of discomfort) and 100 (high stress level) with an increase after noxious stimulation. We will investigate the relationship between the SPI during emergence period and the pediatric assessment of emergence delirium (PAED) score.

SECONDARY OUTCOMES:
The sensitivity and specificity of the SPI in detecting the emergence delirium | Observation from approximately 1 hour after the end of operation
  Receiver operating characteristics (ROC) curves and the associated areas under the curves (AUC) were computed to characterize the sensitivity and specificity of the SPI in detecting a pediatric emergence at different PAED scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Daegu Catholic Medical Center, Daegu, South Korea